CLINICAL TRIAL: NCT04876222
Title: Direct or Subacute Coronary Angiography in Patients With Out of Hospital Cardiac Arrest Without Coma. A Prospective Randomized Study.
Brief Title: Direct or Subacute Coronary Angiography in Patients With Out of Hospital Cardiac Arrest Without Coma.
Acronym: DISCO-noCOMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Aalborg University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, Principal investigator, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DISCO-no-COMA
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Angiography; Percutaneous Coronary Intervention; Coma
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Coma

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute CAG (Active Comparator): The patient is triaged directly to the catheterization laboratory for acute evaluation including ECHO, acute CAG and PCI if indicated according to guidelines.
  Interventions: Procedure: Acute CAG
- Subacute CAG (No Intervention): The patient is triaged to the coronary care unit (CCU) for rhythm surveillance, and additional diagnostics, and in case there is found indication for CAG, it is planned for the coming day in daytime (12-24 hours after cardiac arrest). Revascularization is performed if indicated according to guidelines.

INTERVENTIONS:
Procedure: Acute CAG — The patient is triaged directly to the catheterization laboratory for acute evaluation including ECHO, acute CAG and PCI if indicated according to guidelines.
  Arms: Acute CAG

SUMMARY:
In patients with Out-of-Hospital Cardiac arrest who achieves Return Of Spontaneous Circulation (ROSC) The investigators want to evaluate whether there is a benefit from acute Angiography compared to subacute (12-24 hours) Angiography

DETAILED DESCRIPTION:
Background: The majority of patients with out-of-hospital cardiac arrest (OHCA) have ischemic heart disease (IHD). If signs of ST-elevation myocardial infarction (STEMI) acute coronary angiography (CAG) and primary percutaneous coronary intervention (PPCI) is recommended. In most cases, patients with OHCA who does not achieve Return Of Spontaneous Circulation (ROSC) are also triaged directly to a tertiary center with the possibility to establish mechanical circulatory support, e.g. Extracorporeal Cardiopulmonary Resuscitation (eCPR) (Figure 1). For the remaining group of patients with OHCA who achieves ROSC and have no signs of STEMI it is unsettled whether there is a benefit of acute CAG.

A large international study (Direct or Subacute COronary angiography in out-of-hospital cardiac arrest - DISCO) from Uppsala, Sweden, will study the role of acute CAG in 1006 patients with OHCA who are comatose after achieving ROSC (2). In the Swedish study they only include comatose patients, and randomize patients to either acute CAG or CAG after 3 days.

Three of four Danish tertiary centers have decided to join the Swedish DISCO-study (From now on named DISCO-MAIN).

However, many OHCA patients are not comatose, and without signs of STEMI, thus not eligible for DISCO-MAIN. The investigators also want to investigate the role of acute CAG in these patients, which is the purpose of the current study, named DISCO-no-COMA (Direct or subacute coronary angiography in patients with out-of-hospital-cardiac arrest who are not comatose). This study will include patients in parallel with the DISCO-MAIN-study. This means that all patients with OHCA who receive ROSC and do not fulfill the criteria for acute CAG (STEMI) can be randomized in either DISCO-MAIN (if comatose) or DISCO-no-COMA (if not comatose).

This means that a patient with OHCA without obvious non-cardiac cause, should be triaged as follows (See figure 1):

1. ROSC not achieved (ongoing CardioPulmonary Resuscitation (CPR)): These patients are triaged directly to the catheterization laboratory with the possibility to establish ECPR treatment (5) and perform CAG/PCI (percutaneous coronary intervention) and implant pacemaker if indicated.
2. Signs of STEMI: These patients are triaged directly for acute CAG according to guidelines (6).
3. ROSC, COMA (Glasgow coma scale <=8), not STEMI: Should be included in the DISCO-MAIN trial.
4. ROSC, Glasgow coma scale >8, not STEMI: Should be included in the DISCO-no-COMA trial.

Purpose:

To randomize non-comatose (Glasgow coma scale >8) OHCA survivors for acute CAG or subacute CAG (after 12-24 hours).

Study period: 1.5.2021 to 1.5.2026.

Centers eligible for participation: Danish and European centers. The investigators will primarily contact centers already participating in the DISCO-MAIN trial. Currently all four Danish Tertiary centers participate and up to 8 centers from the Netherlands have agreed to participate.

Patients are randomized to:

Group A: Acute CAG: The patient is triaged directly to the catheterization laboratory for acute evaluation including Echocardiography (ECHO), acute CAG and PCI if indicated according to guidelines.

Group B: Subacute CAG: The patient is triaged to the coronary care unit (CCU) for rhythm surveillance, and additional diagnostics, and in case there is found indication for CAG, it is planned for the coming day in daytime (12-24 hours after cardiac arrest). Revascularization is performed if indicated according to guidelines.

Revascularization in group A and B:

The goal is to perform revascularization of the culprit lesion. Additional lesions will be scheduled for an elective procedure, typically after 3-4 weeks. If Coronary Artery Bypass Grafting (CABG) is indicated, it will be scheduled according to the centers local routine.

Cross-over:

A patient randomized to group B will be scheduled for acute CAG if:

1. Signs of STEMI (acute CAG mandatory).
2. Persistent hemodynamic instability of more than 1 hour after randomization, defined as: need of increased dose of vasopressor/inotropic, low Left ventricular ejection fraction (LVEF), no clearance of lactate (Acute CAG should be considered)
3. Recurrent cardiac arrest (Acute CAG should be considered)
4. Patients who after admission is judged to have NSTEMI can cross-over to acute CAG if they are not stabilized medically.

Statistics: Data is analysed according to intention-to-treat. Continuous data will be presented as mean ± standard deviation, and comparison made using t-test if normally distributed. Non-normal distributed data will be presented as median [interquartile range], and compared using Mann Whitney U-test. Categorical variables are compared using Fischers exact test or Chi square test as appropriate, and presented as numbers and per centages. Significans level is p< 0.05 (two-sided).

Data management: Data will be collected and stored according to the Danish Privacy Law. The E-CRF (Electronic Case Report Form) is computer-based (TrialPartner). Patient and procedure information will be entered in the E-CRF by the study nurses at each site. Date is also collected from the CPR-register, the Danish National Patient Register (LPR-register), as well as the invasive registries covering procedure related data for all patients who have CAG or PCI performed. TrialPartner is approved according to Danish regulative, and all access and data-entry are logged. When the study is finalized and data from the various registries have been merged, the personal identification number is removed, and all cases are assigned a key. A separate key file is store. Data is then made anonymous.

Inclusion of patients and consent:

All patients with OHCA without obvious non-cardiac cause are triaged to the invasive centers. The physician on call ensures that any patient with STEMI or ongoing CPR are triaged directly to the catheterization laboratory. Remaining patients are included in the DISCO-MAIN study if comatose. Non-comatose patients are included in the present DISCO-no-COMA study. They are included according to the paragraph "Research in acute situations", and are randomized when they are still in the prehospital phase if possible, en route to the hospital. After arrival to the hospital, the investigators will inform the patient further, to achieve written informed consent also.

Ethical aspects:

The investigators believe it is legitimate to randomize patients to acute or subacute CAG because Denmark nationally have centers that adhere to both strategies, and it is uncertain whether there is a benefit from acute CAG in OHCA patients who have achieved ROSC and are without signs of obvious STEMI.

Furthermore, there are clear recommendations when to cross-over if randomized to a conservative strategy.

Withdrawal from the study: The patients can at any point, and without any reason, decide not to participate in the study. The patient will be asked if data collected from randomization and until withdrawal may be used. Otherwise data will be deleted. Reason for withdrawal, and the patient's decision whether data can be used or not, will be filled in the electronic health record.

Biobank / biological material: No biobank is collected at present.

Blinding: The study is not blinded, which seems impossible to do.

Personal data:

The national Privacy Law will be followed. The trial will be filed to the Central Denmark Region (Instead of the Danish Data Protection Agency, according to current practice), to the Ethical Committee in the Central Denmark Region and to Clinicaltrials.gov. The National Board of Health will be aplied for access to data from the CPR-register and the National Patient Register.

Access to data: Data will be stored in TrialPartner. Any access or attempt to access will be logged. Investigator/institution will grant access for monitoring and audit also from the ethical committee. Investigator will be responsible and ensure that any patient has given written consent, or a deputy consent has been achieved according to the rules for research in acute situations.

Endpoint committee: An endpoint committee will be established consisting of a cardiologist and an anesthesiologist who validates all clinical endpoints, and establish the final diagnosis (cause of cardiac arrest) for the patient. They will have access to all study material as well as information from patient health records if necessary.

Coordinating center: The research department at the Department of cardiology, Aarhus University hospital, will be the coordinating center, and responsible for establishing the eCRF, collecting data, coordinating safety and endpoint committee meetings, and publish data.

Monitoring: Aarhus University hospital will be responsible for trial monitoring. Study nurses will visit each hospital when initiating the trial, and then approximately two times during the study. The monitoring visits will as in the DISCO-MAIN trial focus on: a) That the study adheres to the protocol, b) that inclusion of patients is according to protocol and inclusion criteria, c) that the correct data is entered in the ECRF, and d) that necessary resources are available locally to perform the study.

Economy: The investigators will apply private funds for support to the study. The responsible physicians will receive no honorarium.

Publications: All results, positive and negative or inconclusive will be published.

Power calculation:

There are limited data on mortality, and risk of recurrent cardiac arrest or cardiogenic shock, in patients without coma who have achieved ROSC after OHCA and just waits for CAG. In previous studies the 30-day mortality was 34% in patients with Acute Myocardial Infarction (AMI) who had Ventricular Tachycardia (VT) or Ventricular Fibrillation (VF) (7), the risk of cardiogenic shock was 9% in patients with VT and 27% in patients with VF (8), and the risk of recurrent cardiac arrest was 7% within 48 hours (8). In the light of competing risks, and in the light of a general reduction in case-fatality during the years, it is assumed that the risk of the combined endpoint (MACE) is approximately 30% within 30 days of randomization. With an alfa of 0.05, and power of 80%, it will be possible to document a difference in MACE of 25% if 1080 patients are included. With an expected drop-out of 10% the aim is to include 1200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed Cardiac Arrest
* ROSC
* CAG possible within 120 minutes
* Glasgow coma scale >8

Exclusion Criteria:

* Age < 18 years
* Obvious non-cardiac cause for the arrest
* Terminal illness
* STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 30-day
  Mortality, cardiogenic shock or recurrent cardiac arrest

SECONDARY OUTCOMES:
Mortality | 30-day and 1-year and 5-year
  All-cause mortality
Cardiogenic shock | 30-day and 1-year
  Lactate>2.5 mmol/l and systolic blood pressure<90 mmHg or need of inotropic
Recurrent cardiac arrest | 30-day and 5-year
  Recurrent cardiac arrest
Revascularization | 30-day and 1-year
  Proportion revascularised with PCI or CABG
Cerebral Performance Category score | 30-day and 6-month
  Cerebral Performance Category (CPC) score. Range 1-5. Lowest number equals best outcome.
modified Ranking Scale score | 30-day and 6-month
  modified Ranking Scale (mRS) score. Range 0-6. Lowest number equals best outcome.
EQ-5D-5L score | 30-day and 6-month
  EQ-5D-5L score
Glasgow Outcome Scale Extended | 6-month
  Glasgow Outcome Scale Extended (GOSE). Range 1-8. Highest number equals best outcome.
Montreal Cognitive Assessment | 6-month
  Montreal Cognitive Assessment (MOCA). Range 0-30. Highest number equals best outcome.
AMPS | 6-month
  AMPS (Assessment of Motor and Process Skills) score. Includes assessment of 16 item motor and 20 item process skills. For each item a score with range 1-4 with. Highest score equals best outome.
ADL-1 score | 6-month
  ADL-1 (Activity of Daily Living) score
Shock from ICD | After randomization and within 30-day and 5-year
  Shock from Implantable Cardiodefibrillator after randomization
AMI | 1-year
  Acute Myocardial Infarction
Readmission with CHF | 1-year
  Readmission with congestive heart failure
Treatment with ICD | 1-year
  Treatment with Implantable Cardiodefibrillator
Bleeding | 30-day
  Drop in Hbg>=1.86 mmol/l or more than 2 units blood
Increase in creatinin | 30-day
  Increase in creatinin more than 100%
Dialysis | 30-day
  Dialysis in patients not previously on dialysis
Vascular surgery | 30-day
  Vascular surgery at access site
Cross-over rate | During admission, 30-day
  Prorportion in subacute group that cross-over to acute angiography before planned
Admission time | 30-day
  Total admission time
MWA index | 1-day and 3-day
  Regional Global Myocardial Work Index assessed by Echo
Renal resistive index | 1-day and 3-day
  Renal restistive index measured by ultrasound to predict renal insuifficiency
Renal and liver flow | 1-day, 3-day, 6-month
  Renal and liver flow measured by ultrasound

CONTACTS AND LOCATIONS:
Locations (7):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Christian Juhl Terkelsen, Aarhus
  - Department of cardiology, Aarhus University Hospital in Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Netherlands (2):
  - Catharina Zeikenhuis, Eindhoven
  - Radboud Universitair Medisch Centrum, Nijmegen